CLINICAL TRIAL: NCT02586831
Title: A Pilot, Safety and Feasibility Trial of Anti-Thymocyte Globulin (ATG), Low Dose Interleukin-2 (IL-2), Adalimumab and Exenatide in the Treatment of New-Onset Type 1 Diabetes
Brief Title: Diabetes Islet Preservation Immune Treatment
Acronym: DIPIT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study withdrawn prior to enrollment due to funding issues
Sponsor: Camillo Ricordi and Jay Skyler (Other)
Collaborators: Diabetes Research Institute Foundation (Other)
Responsible Party: Sponsor-Investigator, Camillo Ricordi and Jay Skyler, Professors, University of Miami Miller School of Medicine and Director/Deputy Director, Diabetes Research Institute, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20150856
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia; Autoimmune Diseases; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Autoimmune Diseases; Diabetes Mellitus | interventions — Antilymphocyte Serum; thymoglobulin; Interleukin-2; aldesleukin; Exenatide; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants in this group will receive Thymoglobulin, Aldesleukin, Adalimumab, and Exenatide over a period of 52 weeks.
  * Anti-Thymocyte Globulin (ATG or Thymoglobulin®) will be administered at a dose of 2.5mg/kg (2 infusions, 0.5 and 2mg/kg) Days 1 and 2
  * Adalimumab (Humira®) will be administered at a dose of 50 mg every month, for 1 year
  * Low-dose Interleukin 2 (Aldesleukin; IL-2 or Proleukin®) will be administered 1 million IU/dose; 5 consecutive days (days 10-14), & then every 2 weeks, for 52 weeks
  * Exenatide (Bydureon®): 2 mg SC weekly up to 52 weeks.
  Interventions: Drug: Anti-Thymocyte Globulin (ATG); Drug: Interleukin 2; Drug: Exenatide; Drug: Adalimumab
- Arm B (Placebo Comparator): Participants in this group will receive the placebos for Thymoglobulin, Aldesleukin, Adalimumab, Exenatide, and Neulasta over a period of 52 weeks.
  Interventions: Other: ATG Placebo; Other: IL-2 Placebo; Other: Adalimumab Placebo; Other: Exenatide Placebo

INTERVENTIONS:
Drug: Anti-Thymocyte Globulin (ATG) — 2.5 mg/kg administered as two divided infusions of 0.5 mg/kg and 2 mg/kg on Days 1 and 2.
  Other Names: Thymoglobulin
  Arms: Arm A
Drug: Interleukin 2 — 1 million IU per dose administered subcutaneously for 5 consecutive days on Days 10-14, and then every two weeks.
  Other Names: Aldesleukin; IL-2 or Proleukin®
  Arms: Arm A
Drug: Exenatide — 2 mg administered subcutaneously weekly for up to 52 weeks.
  Other Names: Bydureon®
  Arms: Arm A
Drug: Adalimumab — 50 mg administered subcutaneously once a month for 1 year.
  Other Names: HUMIRA®
  Arms: Arm A
Other: ATG Placebo — ATG placebo mimicking Thymoglobulin administered intravenously.
  Arms: Arm B
Other: IL-2 Placebo — IL-2 placebo mimicking Aldesleukin administered subcutaneously.
  Arms: Arm B
Other: Adalimumab Placebo — Placebo mimicking Adalimumab administered subcutaneously.
  Arms: Arm B
Other: Exenatide Placebo — Placebo mimicking Exenatide administered subcutaneously.
  Arms: Arm B

SUMMARY:
To assess whether there is a difference in endogenous insulin secretion, measured as stimulated C-peptide secretion (area under the curve during a 4-hour mixed meal tolerance test), at the 1 year visit, for study subjects receiving combinational therapy versus those receiving placebo. The study will also examine the effect of the proposed treatments on immunological outcomes, specifically proportion of regulatory T cells at the 1 year visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible to participate in this study:

  1. Subject must be able to understand and provide informed consent.
  2. Males and females, 18-35 years of age.
  3. New onset T1D for no longer than 120 days at the time of randomization.
  4. Affected by T1D, according to ADA standard criteria, and confirmed by positivity of at least one T1D-associated autoantibody, to GAD65, IA-2, ZnT8, or insulin autoantibodies (if patient has been treated with insulin for less than 2 weeks).
  5. Being on insulin therapy.
  6. Stimulated C-peptide peak level >0.2 nmol/L at the baseline 1 visit MMTT.
  7. Female subjects of childbearing potential must have a negative pregnancy test upon study entry.
  8. Female (and male) subjects with reproductive potential must agree to use two FDA approved methods of birth control for the entire duration of the study.
  9. Adequate venous access to support study required blood draws.

Exclusion Criteria:

* Potential participants must not meet any of the following exclusion criteria:

  1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
  2. BMI>30 Kg/m2.
  3. Contra-indications to ATG, GCSF, exenatide, etanercept and IL-2 (as per package insert, e.g., knowledge of hypersensitivity to drugs or its excipients).
  4. Uncompensated heart failure, fluid overload, myocardial infarction or liver disease or severe impairment of a vital organ within the last 6 weeks before enrollment.
  5. Any of the following laboratory findings: hemoglobin <10.0 g/dL; leukocytes <3,000/μL; neutrophils <1,500/μL; lymphocytes <800/μL; platelets <100,000/μL.
  6. Any sign or diagnosis of significant chronic active infection (e.g., hepatitis, tuberculosis, EBV, or CMV), or screening laboratory evidence consistent with a significant chronic active infection (such as positive for HIV, IGRA test for TB, or hepatitis B-C).
  7. Ongoing acute infections, e.g., acute respiratory tract urinary tract, or gastrointestinal tract infections.
  8. Ongoing or anticipated use of diabetes medications other than insulin.
  9. Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within prior 7 days of screening.
  10. Current or prior use of immunomodulators or systemic steroids in the last 2 months that could potentially affect diabetes or immunologic status.
  11. Recent recipient of any licensed or investigational live attenuated vaccine(s) within 6 weeks of randomization.
  12. Use of investigational drugs within 3 months of participation.
  13. Concomitant therapy with immunosuppressive drugs, immunomodulators, or cytotoxic agents, or previous therapy less than 3 months from randomization.
  14. History or diagnosis of malignancy. Any history of gastroparesis or other severe gastrointestinal disease, pancreatitis, thyroid nodules or malignancy with the exception of a history of localized basal cell carcinoma.
  15. Presence of an allograft.
  16. AST, ALT or Alkaline Phosphatase >2 times upper limit of normal or total bilirubin >1.5 times upper limit of normal.
  17. Current, diagnosed, mental illness or current, diagnosed or self-reported drug or alcohol abuse; or any situation that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
  18. Pregnancy or ongoing breastfeeding for women; unwillingness or inability of both females and males of childbearing age to use a reliable and effective form of contraception, for the entire duration of the study.
  19. Past or current medical problems, or findings from physical examination, or laboratory testing, that are not listed above which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Simulated C-peptide AUC | 1 Year Visit
  Endogenous insulin secretion as measured as stimulated C-peptide section Area Under the Curve (AUC) during a 4 hour mixed meal tolerance test (MMTT)
Proportion of regulatory T cells | 1 Year Visit
  As measured from blood samples

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c) levels | Up to 18 months
  Measure of glycemic control as evaluated by HbA1c levels from blood samples
Insulin dose | Up to 18 months
  Measure of glycemic control as evaluated by insulin dose
Mean daily plasma glucose levels | Up to 18 months
  Measure of glycemic control as evaluated by the mean daily plasma glucose levels from blood samples
Incidence of immune response adverse events | Up to 18 months
  Incidence of immune response adverse events as assessed by treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, M.D., Principal Investigator — Diabetes Research Institute, University of Miami

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skyler JS. Prevention and reversal of type 1 diabetes--past challenges and future opportunities. Diabetes Care. 2015 Jun;38(6):997-1007. doi: 10.2337/dc15-0349. PMID 25998292
- [Background] Skyler JS, Ricordi C. Stopping type 1 diabetes: attempts to prevent or cure type 1 diabetes in man. Diabetes. 2011 Jan;60(1):1-8. doi: 10.2337/db10-1114. No abstract available. PMID 21193733